CLINICAL TRIAL: NCT02407041
Title: A Single-Center, Open-Label Phase 2a Clinical Trial to Evaluate the Safety and Efficacy of GR-MD-02 for the Treatment of Patients With Moderate to Severe Plaque Psoriasis
Brief Title: An Open-Label, Phase 2a Study to Evaluate Safety and Efficacy of GR-MD-02 for Treatment of Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galectin Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GT-030
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Results first posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — belapectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GR-MD-02 (Experimental): active arm
  Interventions: Drug: GR-MD-02

INTERVENTIONS:
Drug: GR-MD-02 — IV infusion
  Other Names: galactoarabino-rhamnogalacturonate

SUMMARY:
Study GT-030 is a phase 2a, single-center, open-label study of subjects with moderate to severe plaque psoriasis

DETAILED DESCRIPTION:
The overall objective is to establish the safety and efficacy of GR-MD-02 in patients with moderate to severe plaque psoriasis.

Primary objective:

The objective is to evaluate the number of patients with moderate to severe plaque psoriasis who have 75% improvement in Psoriasis Activity Severity Index (PASI-75) following 12 weeks of therapy with GR-MD-02

Secondary objectives:

* To determine the PASI-50 and PASI-100 scores in patients with moderate to severe plaque psoriasis following the first 12 weeks of therapy with GR-MD-02
* To determine the PASI-50, PASI-75, and PASI-100 scores in patients with moderate to severe plaque psoriasis following an additional 12 weeks of therapy (total 24 weeks) with GR-MD-02
* To determine the durability of response to therapy in responders over a one year period following the end of therapy
* To determine whether there is any change in disease status of patients who also have psoriatic arthritis
* To determine the incidence of adverse events and vital sign and laboratory abnormalities during study treatment

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all of the following criteria to be enrolled in this study:

1. Is capable of understanding the written informed consent, provides signed and witnessed written informed consent, and agrees to comply with protocol requirements.
2. Is between the ages of 18 and 75 years.
3. Has biopsy proven psoriasis and active moderate to severe plaque psoriasis with a PASI of ≥ 12 and at least 10% of involved body surface area.
4. The patient is not pregnant and must have a negative pregnancy test prior to start of the study. Post-menopausal women must have been amenorrheic for at least 12 months to be considered of non-child-bearing potential.
5. Sexually active men or women of childbearing potential must agree to use effective means of contraception throughout their participation in this study and for 90 days after discontinuation of study medication.
6. Lactating females must agree to discontinue nursing before the start of study treatment and refrain from nursing until 90 days after discontinuation of study medication.
7. Male subjects must refrain from sperm donation throughout the study period and for a period of 90 days following the last dose of study drug.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Any medical illness that is not stable on therapy
2. Use of any biologic medication for psoriasis within 6 months
3. Use of or non-biological systemic therapy to include: methotrexate, oral retinoids, phototherapy/PUVA, cyclosporine, or any other cytotoxic or immunosuppressive medication within 4 weeks of start of study
4. Topical treatment that is likely to impact signs and symptoms of psoriasis, in the opinion of the Principal Investigator, within 2 weeks of the start of the study
5. Prior exposure to GR-MD-02
6. Known positivity for Human Immunodeficiency Virus (HIV) infection
7. Any patient who had major surgery within 8 weeks of Day 1, significant traumatic injury, or anticipation of need for major surgical procedure during the study.
8. Has a history of alcohol/drug abuse.
9. Any patient who has clinically significant and uncontrolled cardiovascular disease (e.g., uncontrolled hypertension, myocardial infarction, unstable angina), New York Heart Association (NYHA) Grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, or Grade II or greater peripheral vascular disease within 12 months prior to Day 1.
10. Any patient with concurrent infection including diagnoses of fever of unknown origin (FUO) (subjects must be afebrile at the start of therapy).
11. History of malignant disease with a recurrence of that disease within 5 years of follow-up except for those that have been curatively treated including basal or squamous cell carcinoma of the skin and in situ carcinoma of the cervix
12. Participation in an investigational new drug (IND) trial in the 30 days before randomization.
13. Clinically significant medical or psychiatric condition considered a high risk for participation in an investigational study.
14. Has donated or lost a significant volume (>450 mL) of blood or plasma within 30 days of the study.
15. Failure to give informed consent
16. Subjects with known allergies to the study drug or any of its excipients.
17. Is an employee or family member of the investigator or study site personnel.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-09; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brooke Army Medical Ctr., San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GR-MD-02
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- GR-MD-02 8 mg/kg: active arm, 8 mg/kg
  GR-MD-02: IV infusion
Arm/Group | GR-MD-02 8 mg/kg
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (19.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With PASI-75, or a 75% Improvement From Baseline in PASI Score
Description: The primary endpoint will be the number of participants with PASI-75, or a 75% improvement from baseline (day 1, prior to first infusion) in PASI score as assessed at the 30 day follow up visit.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | GR-MD-02 8 mg/kg
Number analyzed (Participants) | 5
Participants | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | GR-MD-02 8 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT02407041/Prot_SAP_000.pdf